CLINICAL TRIAL: NCT07374471
Title: A Phase 1b/2a, Multicenter, Double-Blind, Placebo-Controlled Study to Evaluate the Safety, Efficacy, and Pharmacokinetics of MB-001 in Participants With Moderately to Severely Active Ulcerative Colitis
Brief Title: A Study of MB-001 in Moderately to Severely Active Ulcerative Colitis
Status: Not yet recruiting | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: Mage Biologics (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: MB-001-102; 2025-524719-35-00 (EU CTIS Number)
Record Dates: First submitted 2026-01-09; First posted 2026-01-28 (Actual); Last update posted 2026-01-28 (Actual); Status verified 2026-01

CONDITIONS: Ulcerative Colitis (UC)
Keywords: Efficacy study; Oral biologic; Ulcerative Colitis; IBD
MeSH Terms: conditions — Colitis, Ulcerative

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- MB-001 capsules (Experimental): oral capsule formulation
  Interventions: Biological: MB-001
- Matching placebo (Placebo Comparator)
  Interventions: Biological: Matching placebo to MB-001

INTERVENTIONS:
Biological: MB-001 — oral capsule formulation
  Arms: MB-001 capsules
Biological: Matching placebo to MB-001 — oral capsule formulation
  Arms: Matching placebo

SUMMARY:
The goal of this clinical trial is to learn if MB-001, an oral biologic, is able to treat patients with ulcerative colitis. Participants will be asked to take MB-001 or a matching placebo once-daily for a period of 12 weeks. Researchers will compare MB-001 to placebo to investigate its effects on clinical symptoms as well as endoscopic and histopathological findings. Patients will be offered open-label extension for another 12 weeks following the double-blind, placebo-controlled part of the study. Participants will keep a daily diary to record their symptoms and will have up to nine clinic visits.

DETAILED DESCRIPTION:
This double-blind, placebo controlled clinical trial is intended to study the effects of oral MB-001 in patients with moderately to severely active ulcerative colitis. The primary objectives of the study are to assess safety and efficacy. Secondary and exploratory endpoints are endoscopic response, histological response, pharmacokinetics, and pharmacodynamic changes compared to baseline.

ELIGIBILITY:
Inclusion Criteria:

* Nonpregnant, nonlactating adults with a diagnosis of UC extending ≥ 15 cm from the anal verge, established at least 3 months prior to Screening by clinical and endoscopic evidence of UC (colonoscopy or flexible sigmoidoscopy) and confirmed by histology.
* Moderately to severely active UC, defined as an mMS of 5 to 9, inclusive, with MES of at least 2 and RB subscore of at least 1.
* At Screening, a colonoscopy will be required if the participant has had extensive colitis or pancolitis of > 8 years duration or left-sided colitis of > 12 years duration but has not had a colonoscopy within 1 year of the initial Screening visit. If the participant has had a colonoscopy within 1 year of the initial Screening date, a flexible sigmoidoscopy may be used instead.
* Demonstrated, in the opinion of the investigator, an inadequate response, loss of response, or intolerance/medical contraindication to at least 1 of the following treatments at doses approved for the treatment of UC:

  * Oral 5-ASA compounds or sulfasalazine
  * Oral corticosteroids (eg, prednisone, budesonide)
  * Immunosuppressants (eg, AZA, 6-MP, MTX)
  * An approved anti-integrin antibody (eg, vedolizumab)
  * An approved anti-IL-12/23 antibody (eg, ustekinumab)
  * An approved anti-IL-23 p19 antibody (eg, risankizumab, guselkumab, or mirikizumab)
  * An approved S1PR modulator (eg, ozanimod or etrasimod) Note: Participants who have had an inadequate response to more than 1 advanced therapy (eg, anti-integrin, anti-IL 12/23, IL-23 p19 antibody, or S1PR modulator) are not eligible (see Exclusion Criterion #15).
* Participant may be receiving a therapeutic dosage of the following drugs:

  * Oral 5-ASA compounds or sulfasalazine, prescribed dose must be stable for at least 2 weeks before Screening endoscopy or stopped at least 2 weeks prior to Screening endoscopy
  * Oral corticosteroids - prednisone (max. 20 mg/day) (or equivalent) or budesonide (max. 9 mg/day) and have been at a stable dose for at least 2 weeks prior to Screening endoscopy or stopped at least 2 weeks prior to Screening endoscopy
  * Immunosuppressants (AZA, 6-MP, MTX) if the prescribed dose has been stable for at least 8 weeks before Screening endoscopy or stopped at least 8 weeks prior to Screening endoscopy
* POCBP:

  1. Is eligible to participate if not pregnant or breastfeeding, and the following conditions apply:

     * Of childbearing potential and using an acceptable contraceptive method during treatment with the IMP and for a minimum until 28 days after the last dose of IMP. The investigator should evaluate the potential or contraceptive method failure (eg, noncompliance, recently initiated) in relationship to the first dose of IMP. AND
     * Must have a negative highly sensitive pregnancy test as required by local regulations within 24 hours before the first dose of IMP,
  2. Must agree not to donate eggs (ova, oocytes) for the purpose of assisted reproduction during the study and for a period of 28 days after receiving the last dose of IMP.
* Able to participate fully in all aspects of this clinical trial. Full comprehension of consent language and informed consent must be obtained from the participant, or the participant's legally acceptable representative.

Exclusion Criteria:

* The following complications:

  * Acute severe ulcerative colitis, defined by at least 6 bloody diarrhea/day AND any 1 of the following criteria: pulse > 90 beats/min, temperature > 37.8°C, hemoglobin < 105 g/l, erythrocyte sedimentation rate > 30 mm/h, or C-reactive protein > 30 mg/l, or in the investigator's opinion, hospitalization for the treatment of UC may be imminent
  * Previous extensive colonic resection (subtotal or total colectomy)
  * Short bowel syndrome
  * Ileostomy, colostomy, ileoanal pouch, fistulae, or known fixed symptomatic stenosis of the intestine
  * Toxic megacolon or recent history (within less than 6 months) of toxic megacolon or bowel perforation
* Diagnosis of CD or the presence or history of a fistula consistent with CD, indeterminate colitis, ischemic colitis, NSAID-induced colitis, idiopathic colitis (ie, colitis not consistent with UC), radiation colitis, microscopic colitis, infectious colitis, colonic mucosal dysplasia, or untreated bile acid malabsorption.
* Primary sclerosing cholangitis with uncontrolled liver function
* Malignancies or history of malignancy within 5 years of Screening (including solid tumors and hematological malignancies), except for adequately treated or completely excised nonmetastatic basal cell carcinoma, squamous cell carcinoma of the skin, or cervical carcinoma in situ.
* History of adenomatous polyps, unless removed.
* History of lymphoproliferative disease, including lymphoma, or signs and symptoms suggestive of possible lymphoproliferative disease, such as lymphadenopathy and/or splenomegaly.
* Class III or IV cardiovascular morbidity.
* Clinically significant abnormal vital signs, physical examination, or 12-lead ECG at Screening or Day 1 (prolonged QTc using Fredericia's formula [> 460 ms for males and > 470 ms for females]), or conditions leading to additional risk for QT prolongation (eg, congenital long-QT syndrome). Participants with electrolyte abnormalities such as hypokalemia and hypomagnesemia that would increase the risk of QT prolongation should be corrected prior to randomization (an ECG may be repeated after electrolyte correction for determining eligibility, if needed).
* History of bleeding disorders (eg, complement disorders, hemophilia, history of uncontrolled bleeding).
* History of any major neurological disorders including stroke, epilepsy, or demyelinating or neurodegenerative disease.
* Increased risk of infectious complications (eg, recent pyogenic infection, any congenital or acquired immunodeficiency [eg, HIV infection], or past organ or stem cell transplantation).
* Systemic or opportunistic infections:

  * A positive diagnostic TB test at Screening (defined as a positive QuantiFERON(R) test). In cases where the QuantiFERON(R) test is indeterminate, the participant may have the test repeated once and if their second test is negative, they will be eligible. In the event a second test is also indeterminate, or QuantiFERON(R) is unavailable, the investigator has the option to perform a PPD skin test. If the PPD reaction is < 5 mm, then the participant is eligible. If the reaction is at least 5 mm, or PPD testing is not done, the participant is not eligible. An exception is made for participants with a history of latent TB who are currently receiving treatment for latent TB, will initiate treatment for latent TB before the first dose of IMP, or have documentation of completing appropriate treatment for latent TB within 3 years prior to the first dose of IMP.
  * A positive test for HBV, as defined by the presence of HBsAg or HBcAb test. Note: If a participant tests negative for HBsAg, but positive for HBcAb, the participant would be considered eligible if no HBV DNA is present, confirmed by HBV DNA polymerase chain reaction reflex testing performed by the central laboratory.
  * A positive test for HCV, as defined by a positive HCVAb test and detectable HCV RNA. Note: Participants who are HCVAb positive without evidence of HCV RNA may be considered eligible (spontaneous viral clearance or previously treated and cured [defined as no evidence of HCV RNA at least 12 weeks prior to randomization]).
  * Evidence of Clostridioides difficile toxin or treatment for C. difficile infection, or other intestinal bacterial pathogen, within 4 weeks prior to Screening.
  * Clinically active cytomegalovirus infection.
  * Any other clinically significant extra-intestinal infection or opportunistic, chronic, or recurring infection within 6 months prior to randomization, including, but not limited to infections requiring IV antibiotics, hospitalization, or prolonged treatment.
  * History of opportunistic infections.
* Autoimmune disorders that may require treatment with immunosuppressant therapy.
* Any of the following laboratory abnormalities during the screening period. If values are initially outside the prescribed limits, the evaluation may be repeated once within the screening period to determine eligibility:

  * Hemoglobin level: < 8.0 g/dL
  * Absolute white blood cell count: < 3.0 x 109/L
  * Absolute lymphocyte count: < 0.5 x 109/L
  * Absolute neutrophil count: < 1.5 x 109/L
  * Platelet count: < 100 x 109/L or > 1200 x 109/L
  * Alanine aminotransferase or aspartate aminotransferase: > 2.5 x ULN
  * Alkaline phosphatase: > 2.5 x ULN
  * Bilirubin: > 1.5 x ULN
* Participants who had an inadequate response to > 1 of the following treatments: vedolizumab, ustekinumab, anti-IL-23 p19 antibodies, or S1PR modulators for UC.
* Participants who had an inadequate response or loss of response to TNF inhibitors or JAK inhibitors.
* Participants taking the following medical therapies for UC:

  * Any biologic therapy (eg, anti-integrins, anti-ILs) within 8 weeks or 5 half-lives (whichever is longer) prior to randomization
  * S1PR modulators within 4 weeks or 5 half-lives (whichever is longer) prior to randomization
  * IV antibiotics within 8 weeks prior to randomization or expected to receive IV antibiotics during the conduct of the study
  * Any rectal therapy for treatment of UC within 2 weeks prior to Screening endoscopy
  * NSAIDs as long-term treatment, defined as use for at least 4 days a week each month (> 100 mg daily or acetaminophen and aspirin > 325 mg daily)
* Any medicinal product, herbal medication, or natural health product which might interfere with peristalsis within 2 weeks prior to randomization.
* Participants unwilling to withhold protocol-prohibited medications during the study.
* Fecal microbiota transplant (includes human microbiota-based therapeutics) within 4 weeks prior to randomization.
* Vaccination with a live or live-attenuated vaccine within 4 weeks prior to randomization, or planned vaccination during conduct of the study.
* Any major surgery, in the investigator's opinion, performed within 8 weeks prior to randomization or planned during the study (ie, any surgical procedure requiring general anesthesia).
* Concurrent or previous participation in another clinical trial and received investigational therapy within 4 weeks or 5 half-lives (whichever is longer) prior to randomization.
* Prior enrolment in the current study and had received IMP.
* History of excessive alcohol or drug abuse that, in the opinion of the investigator, may interfere with the participant's ability to comply with the study procedures.
* Known or suspected allergy, hypersensitivity or intolerance to the IMP or its' excipients.
* Participant is performing mandatory military service, deprived of liberty, in a residential care institution, or due to a judicial decision cannot take part in a clinical study.
* Participant is an immediate family member, study site employee, or is in a dependent relationship with a study site employee who is involved in the conduct of this study (eg, spouse, parent, child, sibling).
* Participant has other severe acute or chronic medical or psychiatric condition or laboratory abnormality that may increase the risk associated with study participation, IMP administration, study participation, or may interfere with the interpretation of study results, as determined by the investigator.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 100 (Estimated)
Dates: Start 2026-04 (Estimated); Primary Completion 2028-07 (Estimated); Study Completion 2028-08 (Estimated)

PRIMARY OUTCOMES:
Incidence of adverse events | From study start until 4 weeks after end of treatment
  All adverse events and serious adverse events will be collected from the signing of the ICF until the safety follow-up visit
Changes in laboratory parameters: Platelet count | Week 12
Changes in laboratory parameter: Hemoglobin | Week 12
Changes in laboratory parameter: Hematocrit | Week 12
Changes in laboratory parameter: Red Blood Cell (RBC) count | Week 12
Changes in laboratory parameter: Prothrombin time | Week 12
Number of participants with abnormal laboratory tests results | Week 12
  Blood urea nitrogen, potassium, creatinine, creatinine phosphokinase, sodium, calcium, glucose, uric acid, AST/serum glutamic-oxaloacetic transaminase, ALT/serum glutamic-pyruvic transaminase, Gamma-glutamyl transferase/transpeptidase, alkaline phosphatase, bilirubin, protein, triglycerides, cholesterol, high-density lipoprotein, low-density lipoprotein
Number of participants with abnormal urinalysis results | Week 12
  Specific gravity, pH, colour, glucose, protein, blood, ketones, bilirubin, urobilinogen, nitrite, leukocyte esterase
Proportion of participants achieving clinical remission | Week 12
  Defined by a modified Mayo Score (mMS) of not more than 2 with a Mayo endoscopic subscore (MES) not more than 1, rectal bleeding (RB) subscore of 0, and stool frequency (SF) subscore not more than 1. The mMS ranges from 0 to 9. Higher values are worse.

SECONDARY OUTCOMES:
Proportion of participants achieving endoscopic improvement | Week 12
  Defined as a May Endoscopy Score (MES) of not more than 1. The MES measures the severity of mucosal inflammation detected during endoscopy and ranges from 0 to 3 with higher values indicating more severe disease.
Proportion of participants achieving endoscopic remission | Week 12
  Defined as a May Endoscopy Score (MES) of 0. The MES measures the severity of mucosal inflammation detected during endoscopy and ranges from 0 to 3 with higher values indicating more severe disease.
Proportion of participants achieving histologic remission | Week 12
  Defined as a Geboes Score of not more than 2B.0. The Geboes sub-score 2B measures the presence of neutrophils in a biopsy sample of the epithelium and ranges from 2B.0 to 2B.3 with higher values indicating more severe disease.
Proportion of participants achieving histologic-endoscopic mucosal improvement | Week 12
  Defined as a Geboes Score not more than 3.1 and Mayo Endoscopy Score (MES) of not more than 1. The Geboes Score 3 measures percent of crypts in a biopsy sample of the epithelium where neutrophils are present and ranges from 3.0 to 3.3 with higher values indicating more severe disease. The MES measures the severity of mucosal inflammation detected during endoscopy and ranges from 0 to 3 with higher values indicating more severe disease.
Proportion of participants achieving mucosal healing | Week 12
  Defined as a Geboes Score of not more than 2B.1 and a Mayo Endoscopy Score (MES) of not more than 1. The Geboes sub-score 2B measures the presence of neutrophils in a biopsy sample of the epithelium and ranges from 2B.0 to 2B.3 with higher values indicating more severe disease. The MES measures the severity of mucosal inflammation detected during endoscopy and ranges from 0 to 3 with higher values indicating more severe disease.

OTHER OUTCOMES:
Area under the plasma concentration-time curve | Week 12
Levels of Anti-Drug Antibodies (ADAs) | Week 12
  Measured by an electrochemiluminescence bridging assay

IPD SHARING:
Plan to Share IPD: Yes
Based on review of a study synopsis and if in line with informed consent criteria
Supporting Information: Study Protocol, ICF
Time Frame: from 2019 onwards
Access Criteria: Researches based on a synopsis as well as evidence of funding